CLINICAL TRIAL: NCT02533947
Title: Effects of Physical Exercise on Cognitive Functions in Patients After Allogeneic Stem Cell Transplantation
Brief Title: Cognition in Allogeneic Stem Cell Transplanted Patients and Sports
Acronym: CaSpo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Deutsche José Carreras Leukämie-Stiftung (DJCLS) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CaSpo; DJCLS R 13/23 (Other Grant/Funding Number: Deutsche José Carreras Leukämie-Stiftung (DJCLS))
Record Dates: First submitted 2015-03-02; First posted 2015-08-27 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Allogeneic Stem Cell Transplantation; Exercise Intervention
Keywords: Allogeneic Stem Cell Transplantation; Hematological Malignancies; Exercise Intervention; Cognitive Function; Fatigue; Randomized Controlled Trial
MeSH Terms: conditions — Hematologic Neoplasms; Fatigue | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise group (Experimental): The exercise program will be developed through a pilot phase with 10 patients prior to the start of the main study.
  Interventions: Behavioral: Exercise
- Control group (Other): A waitlist control group will get the intervention after 7 month of treatment as usual.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Exercise — The intervention consists of an individually tailored supervised exercise program with aerobic, strength and coordinative components.
  Arms: Exercise group
Behavioral: Control — A waitlist control group will get the intervention after 7 month of treatment as usual.
  Arms: Control group

SUMMARY:
Studies suggest that patients with hematological malignancies undergoing allogeneic hematopoietic stem cell transplantation (HSCT) are at risk for cognitive decline and long-term cognitive dysfunction. To address this issue, a randomized controlled intervention trial on the effect of physical exercise on cognition is conducted. In addition, the impact on psychological and physical health outcomes is evaluated. Results may benefit patients who suffer from disease- or treatment-associated cognitive change.

DETAILED DESCRIPTION:
Studies suggest that patients with hematological malignancies undergoing allogeneic hematopoietic stem cell transplantation (HSCT) are at risk for cognitive decline and long-term cognitive dysfunction. To address this issue, a randomized controlled intervention trial on the effect of physical exercise on cognition is conducted. In addition, the impact on psychological and physical health outcomes such as depression, fatigue, health-related quality of life and physical fitness is evaluated. A healthy control group matched to the patients on age, gender, and education will be included to both control for practice effects on neuropsychological measures and allow additional comparisons on self-report measures. The healthy control group will undergo neuropsychological testing and questionnaire survey at baseline and 4 months. Demographic data will be collected from all study participants at baseline. Medical data will be collected from patients at all time points. Results may benefit patients who suffer from disease- or treatment-associated cognitive change.

ELIGIBILITY:
Patients:

Inclusion Criteria:

* hematological malignancy (AML, ALL, MDS, OMF, CML, MM, NHL, Hodgkin, AA)
* 3 to 6 months after allogeneic HSCT
* ≥ 18 years of age at time of transplantation
* German as mother tongue
* regular follow-up visits at the transplantation center during the first year after transplantation

Exclusion Criteria:

* > 75 years of age at time of transplantation
* relapse/progress
* thrombocyte count ≤ 50 G/l
* GvHD with lung involvement
* compromised lung function (patients who need oxygen)
* compromised cardiovascular function (< 10-m walk)
* florid infection
* immobility
* neurological disease
* severe psychiatric disease
* regular intake of psychoactive drugs or substance abuse
* uncontrolled diabetes
* high fracture risk
* impaired vision and/or hearing

Healthy controls (matched for age, gender, and education):

Inclusion Criteria:

* ≥ 18 years of age at time of enrolment
* German as mother tongue
* residence in the area of the transplantation center or family members/friends accompanying the patients to clinical follow-up visits

Exclusion Criteria:

* > 75 years of age at time of enrolment
* hematological malignancy
* solid tumour disease
* neurological disease
* severe psychiatric disease
* regular intake of psychoactive drugs or substance abuse
* impaired vision and/or hearing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-06; Primary Completion 2019-05 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive functioning as assessed by Change in total z-score | Baseline and 4 months
  Change in total z-score derived from a neuropsychological test battery (TMT-A, TMT-B, subtests Alertness, Sustained Attention and Flexibility from the German TAP, German Version of the Rey Auditory Verbal Learning Test, Digit Span from the WAIS-IV, German Version of the COWA, Tower of London).

SECONDARY OUTCOMES:
Change in cognitive functioning as assessed by Change in total z-score | Baseline and 7 months
  Change in total z-score derived from a neuropsychological test battery (TMT-A, TMT-B, subtests Alertness, Sustained Attention and Flexibility from the German TAP, German Version of the Rey Auditory Verbal Learning Test, Digit Span from the WAIS-IV, German Version of the COWA, Tower of London).
Change in self-reported cognitive functioning as assessed by Change in scale sum score (composite score) of the FEDA and FLei questionnaires | Baseline, 4 months, 7 months
  Change in scale sum score of the FEDA and FLei questionnaires measuring self-perceived attentional (FEDA scale 1: Distractibility and Retardation in Mental Processes, FEDA scale 2: Fatigue and Retardation in Activities of Daily Living, FEDA scale 3: Decrease in Drive), memory (FLei scale memory), and executive dysfunctions (FLei scale executive function).
Change in fine-motor function | Baseline, 4 months, 7 months
  Change in z-score derived from the GPT dominant hand
Change in physical fitness (muscle strength) | Baseline, 4 months, 7 months
  Measured with M. quadriceps isometric strength test, one 10-sec trial on each leg (change in mean strength value)
Change in physical ability/capability (walking ability) | Baseline, 4 months, 7 months
  Measured with the 6-min walk test (change in walk distance in meters)
Change in physical activity (intensity) | Baseline, 7 months
  Measured with accelerometry, 1-week period (change in metabolic equivalent task [MET] values)
Change in self-reported physical activity | Baseline, 4 months, 7 months
  Measured with the EPIC Physical Activity Questionnaire
Change in immunological functions | Baseline, 4 months, 7 months
  Severity of GvHD
Change in health-related quality of life | Baseline, 4 months, 7 months
  Measured with the EORTC QLQ-C30 (change in global health status / QoL scale)
Change in fatigue | Baseline, 4 months, 7 months
  Measured with the MFI-20 (change in total score)
Change in anxiety | Baseline, 4 months, 7 months
  Measured with the HADS subscale anxiety (change in subscale score)
Change in depressive symptoms | Baseline, 4 months, 7 months
  Measured with the HADS subscale depression (change in subscale score)
Change in fear of cancer recurrence | Baseline, 4 months, 7 months
  Measured with the PA-F12 (change in sum score)

OTHER OUTCOMES:
Intentional behaviour related to physical activity | 4 months, 7 months
  Measured with the stage of change component of the transtheoretical model
Self-efficacy towards physical exercise | 4 months, 7 months
  Measured with three items (Fuchs, 2008)
Situational barriers for physical exercise | 4 months, 7 months
  Measured with the scale on situational barriers (13 items, Krämer & Fuchs, 2010)
Grip strength | Baseline, 4 months, 7 months
  Measured with a handgrip dynamometer
Inflammation | Baseline, 4 months, 7 months
  High-sensitivity CRP derived from routine blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Karl-Heinz Schulz, Prof.Dr.Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany